CLINICAL TRIAL: NCT05910541
Title: The Efficacy of Multisession Mindful Breathing in Symptom Reduction Among Patients: A Randomised Controlled Trial
Brief Title: The Efficacy of Multisession Mindful Breathing in Symptom Reduction Among Patients With Advanced Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Malaysia Sarawak (Other)
Collaborators: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MREC No. 20191125-8042
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Advanced Cancer
Keywords: mindful breathing, multisession, advanced cancers
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients will receive standard care plus daily sessions of 30-minute mindful breathing for four consecutive days
  Interventions: Behavioral: Mindful breathing; Other: Standard care (control)
- Control (Sham Comparator): Patients will only receive standard care.
  Interventions: Other: Standard care (control)

INTERVENTIONS:
Behavioral: Mindful breathing — 30 minutes of mindful breathing session for 4 consecutive days, guided by investigators in addition to standard care.
  Arms: Intervention
Other: Standard care (control) — Standard care such as pain control, oxygen supplement.

SUMMARY:
The goal of this clinical trial is to determine the efficacy of multisession mindful breathing in reducing symptoms among patients with advanced cancer. Adult patients with advanced cancer will be assessed using Edmonton Symptom Assessment System (ESAS) scoring system. Patients who scored ≥4 in at least two or more components in ESAS will be recruited and randomly assigned to either 4 daily-session of 30-minute mindful breathing and standard care or standard care alone.

DETAILED DESCRIPTION:
Patients with advanced cancer admitted to the medical and surgical wards of UMMC were consecutively approached to screen for eligibility. The 30-minute mindful breathing of the intervention group was guided by similar investigators for four consecutive days. These investigators were medical doctors who had been trained by the primary investigators - a palliative care physician and a certified mindfulness trainer. Each session used different scripts and was conducted in the languages that were preferred by the patients (such as Malay, English, or Mandarin). Briefly, patients were primed with knowledge of the gist of each script before being instructed to relax their bodies, close their eyes, pay attention to their breathing, and follow the guidance given. If they noticed any distractions, they were told to redirect their attention back to their breathing. Patients in the control group only received standard care and were assessed at the same time of the day by similar investigators for four consecutive days. Patients were allowed to continue their usual activities during each session.

ELIGIBILITY:
Inclusion Criteria:

* ongoing stage IIII-IV cancer, and a score of four or more in at least two components

Exclusion Criteria:

* impaired cognition or conscious level, as well as psychiatric illnesses that prevent them from giving informed consent or participating fully in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Total score of ESAS | 30 muinutes
  Assessment of efficacy of multisession 30 minutes mindful breathing on the total score of ESAS

SECONDARY OUTCOMES:
Individual score of the ten symptoms in ESAS | 30 minutes
  Assessment of efficacy of the multisession 30 minutes mindful breathing on the individual score of the 10 symptoms in ESAS.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Leh Ching Ng, MD, Principal Investigator — University Malaysia Sarawak
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang VT, Hwang SS, Feuerman M. Validation of the Edmonton Symptom Assessment Scale. Cancer. 2000 May 1;88(9):2164-71. doi: 10.1002/(sici)1097-0142(20000501)88:93.0.co;2-5. PMID 10813730
- [Result] Bruera E, Kuehn N, Miller MJ, Selmser P, Macmillan K. The Edmonton Symptom Assessment System (ESAS): a simple method for the assessment of palliative care patients. J Palliat Care. 1991 Summer;7(2):6-9. PMID 1714502
- [Derived] Tung YZ, Ng DLC, Lai NZ, Ang CM, Lim PK, Zainuddin SI, Lam CL, Loh EC, Chai CS, Tan SB. Symptom reduction in advanced cancer from multi-session mindful breathing: randomised controlled study. BMJ Support Palliat Care. 2025 Feb 18:spcare-2024-005086. doi: 10.1136/spcare-2024-005086. Online ahead of print. PMID 39965903